CLINICAL TRIAL: NCT06604598
Title: The Effect of NSAID Steroid Therapy for PGE2 Level and Analgesia After Percutaneous Nephrolithotomy Surgery, a Double Blinded Randomised Controlled Trial
Brief Title: The Effect of NSAID Steroid Therapy for PGE2 Level and Analgesia After Percutaneous Nephrolithotomy Surgery
Acronym: BUPARDEX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitas Jenderal Soedirman (Other)
Responsible Party: Principal Investigator, Erni Noviani, Principal Investigator Department Anesthesiology and Intensive Therapy, Universitas Jenderal Soedirman
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUPARDEX
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Percutaneous Nephrolithotomy (PCNL); Postoperative Pain
Keywords: steroid; PGE2; analgesia; percutaneous nephrolithotomy; NSAID; postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Intervention Model Description: BUPARDEX (iBUprofen, PARacetamol, DEXamethasone) is a parallel 3-group, blinded, randomized controlled trial. Participants were randomized using random generator application, and divided to 3 groups in a 1:1:1 ratio. Ibuprofen (Peinlos) 400 mg iv, Paracetamol (Bernofarm) 1 gr iv, dexamethasone (Phapros) 5 mg iv will give within IBU-PCT-DEX intervention. Ibuprofen (Peinlos) 400 mg iv; Paracetamol (Bernofarm) 1 gr iv; and placebo (normal saline alike dexamethasone) will give within the IBU-PCT-placebo intervention. Paracetamol (Bernofarm) 1 gr iv; placebo (normal saline alike paracetamol); placebo (normal saline alike dexamethasone) will give within PCT-placebo-placebo intervention. All drugs manufactured by Indonesia. The study was conducted after obtaining an ethical clearance from the Medical Research Ethics Commission, Faculty of Medicine, Universitas Jenderal Soedirman (No. 052/KEPK/PE/VII/2024). Participant, care provider, investigator, outcome assessor will be blind during trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- PCT-placebo-placebo (Active Comparator): Paracetamol (Bernofarm) 1 gr iv; placebo (normal saline alike paracetamol); placebo (normal saline alike dexamethasone) will be given two times administration, interval 8 hour, within the PCT-placebo intervention.
  Interventions: Drug: PCT-placebo-placebo
- IBU-PCT-placebo (Active Comparator): Ibuprofen (Peinlos) 400 mg iv; Paracetamol (Bernofarm) 1 gr iv; and placebo (normal saline alike dexamethasone) will be given two times administration, interval 8 hour, within the IBU-PCT-placebo intervention.
  Interventions: Drug: IBU-PCT-placebo
- IBU-PCT-DEX (Experimental): Ibuprofen (Peinlos) 400 mg iv, Paracetamol (Bernofarm) 1 gr iv, dexamethasone (Phapros) 5 mg iv will be given two times administration, interval 8 hour, within IBU-PCT-DEX intervention.
  Interventions: Drug: IBU-PCT-DEX

INTERVENTIONS:
Drug: IBU-PCT-DEX — Ibuprofen (Peinlos) 2x400 mg iv, Paracetamol (Bernofarm) 2x1 gr iv, dexamethasone (Phapros) 2x5 mg iv will be given with interval 8 hour, within the IBU-PCT-DEX intervention.
  Other Names: Ibuprofen+paracetamol+dexamethasone
  Arms: IBU-PCT-DEX
Drug: IBU-PCT-placebo — Ibuprofen (Peinlos) 2x400 mg iv, Paracetamol (Bernofarm) 2x1 gr iv, and 2xplacebo (normal saline alike dexamethasone) will be given with interval 8 hour, within the IBU-PCT-placebo intervention
  Other Names: ibuprofen+paracetamol+placebo
  Arms: IBU-PCT-placebo
Drug: PCT-placebo-placebo — Paracetamol (Bernofarm) 2x1 gr iv, 2xplacebo (normal saline alike paracetamol), 2xplacebo (normal saline alike dexamethasone) will be given with interval 8 hour, within the PCT-placebo-placebo intervention.
  Arms: PCT-placebo-placebo

SUMMARY:
The goal of this clinical trial is to learn if combination of NSAID-steroid can decrease the PGE2 level and postoperative pain after percutaneous nephrolithotomy surgery. It will also learn about the side effects of combination of those drugs. The main questions it aims to answer are:

Does combination of NSAID steroid can lower the PGE2 level and NRS score after percutaneous nephrolithotomy surgery? What side effect do participants have when taking combination of NSAID-steroid after percutaneous nephrolithotomy surgery? Researchers will compare Group IBU-PCT-DEX (ibuprofen -paracetamol-dexamethasone), Group IBU-PCT-placebo (ibuprofen-paracetamol-placebo), and Group PCT-placebo-placebo (paracetamol-placebo-placebo) to see the difference level of PGE2 and NRS score after percutaneous nephrolithotomy surgery.

Participants will:

Receive drug intravenously according to group allocation, every 8 hours Report the side effects when taking medication during trial

DETAILED DESCRIPTION:
Our study aim to investigate the effect of NSAID steroid therapy to PGE2 level and analgesia after percutaneous nephrolithotomy surgery. This study is a double blind randomized controlled trial at a primary health care center in Purwokerto, Indonesia. This trial involved 45 patient who underwent elective percutaneous nephrolithotomy surgery who met the inclusion and exclusion criteria. Patient was randomized and divided into three groups. Each group consisted of 15 patients. Ibuprofen 2x400 mg iv + paracetamol 2x1 gr iv + dexamethasone 2x5 mg iv will be given within the IBU-PCT-DEX intervention. Ibuprofen 2x400 mg iv + paracetamol 2x1gr iv + 2xplacebo (normal saline alike dexamethasone) iv will be given within the IBU-PCT-placebo intervention. Paracetamol 2x1 gr iv + 2xplacebo (normal saline alike ibuprofen) + 2xplacebo (normal saline alike dexamethasone) will be given within the PCT-placebo-placebo intervention. The analgesics were given during surgery and 8 hours after first drug administration. Plasma level of PGE2 will be measured with ELISA. and analgesia will be measured using numeric rating scale (NRS) an hour after two times drug administration. Primary outcome was PGE2 level and NRS score after percutaneous nephrolithotomy among three group of comparison. Secondary outcome was the side effect of analgesic.

ELIGIBILITY:
Inclusion Criteria:

1. Elective, percutaneous nephrolithotomy surgery
2. Age ≥ 18 years to ≤ 70 years
3. Body mass index (BMI) > 18 kg/m2 to < 40 kg/m2
4. American Society of Anesthesiologists (ASA) Physical Status Classification System 1-3.
5. Written informed consent to participate in the trial.

Exclusion Criteria:

1. Patients with allergy to ibuprofen, paracetamol, and dexamethasone
2. Patients with uncontrolled diabetes mellitus
3. Patients with previous history of alcohol or drug abuse
4. Patients who unconscious
5. Patients with neurological disorders
6. Patients with cognitive impairment
7. Patients who incapable of communication
8. Patients with daily use of systemic glucocorticoids within 3 months prior to surgery
9. Patients with daily use of high-dose opioid (tramadol 150 mg/day or morphine >30 mg/day orally) or use transdermal opioid
10. Patients who are contraindicated to ibuprofen or paracetamol, include a history of peptic ulcers, renal failure (glomerular filtration rate <60 ml/kg/1.73 m2), heart failure, severe liver dysfunction, thrombocytopenia <100,000/L.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
NRS Score | from enrollment to the end of treatment at 5 weeks
  NRS score will be measured an hour after two times drug administration. The value scale from 0 to 10. Higher scores mean outcome worse.
PGE2 level | from enrollment to the end of treatment at 5 weeks
  PGE2 level will be measured by ELISA elabscience kit. PGE2 level will be measured an hour after two times drug administration, using plasma sample. The result is displayed in pg/ml (numeric scale)

SECONDARY OUTCOMES:
The side effects | from enrollment to the end of treatment at 5 weeks
  The side effects of trial medication to participants including nausea, vomiting, epigastric pain, allergy, and no side effect. Data will be collected after two times drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: M. Mukhlis Rudi Prihatno, Study Director — Universitas Jenderal Soedirman
Locations (1):
- Margono Soekarjo Hospital, Banyumas, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
IPD is privacy according to our ethical research committee

REFERENCES:
- [Background] Momesso GAC, Grossi-Oliveira GA, Silva WPP, Akira R, Chiba F, Polo TOB, de Lima Neto TJ, Rios BR, Bassi APF, Sumida DH, Han M, Miloro M, Faverani LP. A triple-blind randomized clinical trial of different associations between dexamethasone and non-steroids anti-inflammatories for preemptive action in third molar extractions. Sci Rep. 2021 Dec 27;11(1):24445. doi: 10.1038/s41598-021-04068-z. PMID 34961782
- See also: study protocol — http://fk.unsoed.ac.id